CLINICAL TRIAL: NCT06595953
Title: Phase II Efficacy Study of Gaze-Contingent Music Therapy Augmentation of CBT for Pediatric Anxiety
Brief Title: Gaze-Contingent Music Therapy Augmentation of CBT for Pediatric Anxiety
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10001937; 001937-M
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-09-18

CONDITIONS: Psychiatric Disorders; Anxiety Disorders
Keywords: Cognitive-behavioral therapy; Attention; Anxiety; Children; Adolescents
MeSH Terms: conditions — Mental Disorders; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active-GCMRT (Active Comparator): In the active form of the therapy, music stops when subjects view negative valence faces.
  Interventions: Behavioral: Gaze-Contingent Music Reward Therapy
- Sham-GCMRT (Sham Comparator): In the control condition, music plays continuously.
  Interventions: Behavioral: Gaze-Contingent Music Reward Therapy

INTERVENTIONS:
Behavioral: Gaze-Contingent Music Reward Therapy — All subjects will receive CBT and will be randomized to either active or control forms of GCMRT. This involves the monitoring of a patient s eye-movements during the free-viewing of computer-displayed matrices of faces expressing various emotions in tandem with the playing of pleasant music. In the active form of the therapy, music stops when subjects view negative valence faces, whereas in the control condition, music plays continuously. Subjects undergo 12 weeks of CBT, where GCMRT is delivered in the last eight weeks of therapy.

SUMMARY:
Background:

Anxiety disorders are becoming more common among children and teenagers. Anxiety can lead to long-term physical and mental problems, such as depression. Treatments for anxiety disorders include medications as well as cognitive behavioral therapy (CBT); CBT is a form of talking therapy. Both approaches work in only about 50 percent of cases. A new approach, called gaze-contingent music reward therapy (GCMRT), may help.

Objective:

To find out whether GCMRT combined with CBT is more effective than CBT alone.

Eligibility:

Children aged 8 to 17 years with separation anxiety disorder; generalized anxiety disorder; or social anxiety disorder. They must be enrolled in protocol 01-M-0192.

Design:

Participants will come to the clinic once a week for 4 weeks for CBT. Sometimes the participant will meet with the doctor alone; sometimes their parent may be present. They will do some computer-based tasks: They may be asked to push a button when a target appears; they may look at pictures of faces while the computer tracks their eye movements. Participants will take questionnaires each week. They will answer questions about their anxiety symptoms, feelings, and behavior.

For the next 8 weeks, participants will participate in both CBT and 1 of 2 types of GCMRT.

GCMRT is a computer-based task. Participants will look at pictures with many faces in them; while they do this, pleasant music will play and stop playing over a 12-minute period.

Participants will have a final visit in week 13. They will take questionnaires. They will do final research tasks. Each visit lasts about 2 hours.

DETAILED DESCRIPTION:
Study Description:

This study compares the efficacy of Gaze-Contingent Music Reward Therapy (GCMRT) and a control form of GCMRT, both added to concurrent therapy. Efficacy will be examined for the severity of clinician-rated anxiety in medication-free children and adolescents with an anxiety disorder. For concurrent therapy, all patients will receive Cognitive Behavioral Therapy (CBT). With this design, efficacy is based on comparison of groups receiving CBT augmented with either active or control forms of GCMRT. A total of 150 patients will be enrolled in the study and will begin CBT therapy for three weeks. By the end of week three, participants will be randomly assigned in a one-to-one ratio to the two forms of GCMRT, which they will receive along with CBT for 9 weeks. From among the 150 patients who enroll in the study, 120 are expected to be randomized to one of the two forms of GCMRT.

Objectives:

Primary Objective: To test the efficacy of Gaze-Contingent Music Reward Therapy (GCMRT) for the augmentation of Cognitive Behavioral Therapy (CBT) treatment for pediatric anxiety disorders.

Secondary Objective: To test for efficacy on secondary outcome measures as well as to test for moderation and mediation of efficacy by measures of attention bias.

Endpoints:

Primary Endpoint: The severity of clinician-rated anxiety, blinded to the GCMRT condition, on the Pediatric Anxiety Rating Scale (PARS).

Secondary Endpoints: Overall treatment response on the clinician-rated Clinician Global Impression scale and rated symptoms of anxiety on the Screen for Child Anxiety Related Disorders (SCARED) scale, as completed by parents and patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Ability of subject and parent to understand the study and the willingness to assent/consent into the study.
2. Males and females; Age 8-17
3. Clinician confirmed diagnosis of ongoing separation anxiety disorder, generalized anxiety disorder, or social anxiety disorder. A clinician will review a KSADS-PL DSM-5 (November 2016) (Kiddie Schedule for Affective Disorders and Schizophrenia for School Aged Children) interview, which will have occurred on Protocol 01-M-0192, to confirm diagnosis
4. Willingness to adhere to 12 weekly in-person sessions of CBT
5. Enrolled in Protocol 01-M-0192
6. Subjects must speak, read and write English to be able to participate
7. All subjects will have IQ>70 as assessed by a WASI or assessment by trained clinical staff which will have occurred under Protocol 01-M-0192

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Current use of any psychotropic medication
2. Ongoing participation in another treatment or intervention study
3. Ongoing mental health treatment outside of NIH
4. Any mental health diagnosis aside from an anxiety disorder as determined by the Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS)
5. Any serious medical conditions
6. Restrictions that preclude in-person attendance of therapy

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Pediatric Anxiety Rating Scale (PARS) | Week 1-13.
  Completed by the clinician.

SECONDARY OUTCOMES:
Clinical Global Impression Scale (CGI) | Week 1-13.
  Completed by the clinician.
Screen for Child Anxiety Related Disorders (SCARED) | Week 1, 4, and 13.
  Completed by parents and patients.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Pine, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001937-M.html